CLINICAL TRIAL: NCT03825237
Title: Sleep Architecture and Factors Associated With Definitive Diagnosis of Sleep Bruxism: a Case-control Study
Brief Title: Sleep Architecture and Factors Associated With Definitive Diagnosis of Sleep Bruxism
Status: Completed | Type: Observational
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Associate Professor, Federal University of Pelotas
Other Study IDs: FUPelotas3
Record Dates: First submitted 2018-11-19; First posted 2019-01-31 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-06

CONDITIONS: Sleep Bruxism, Adult
Keywords: diagnostic; polysomnography; sleep architecture; sleep bruxism
MeSH Terms: conditions — Sleep Bruxism; Disease | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With sleep bruxism by polysomnography: Adults (20 to 60 years) and elderly (> 60 years), (WHO-World Health Organization, 2015) who had undergone polysomnography (PSG) from January 2015 to December 2017 were assessed. All self-reports and PSG exams were included and reviewed. The participants were excluded if they presented with a history of neurological or degenerative disorders, and any objection to take the polysomnography test.
  Interventions: Diagnostic Test: Polysomnography
- Without sleep bruxism by polysomnography: Adults (20 to 60 years) and elderly (> 60 years), (WHO-World Health Organization, 2015) who had undergone polysomnography (PSG) from January 2015 to December 2017 were assessed. All self-reports and PSG exams were included and reviewed. The participants were excluded if they presented with a history of neurological or degenerative disorders, and any objection to take the polysomnography test.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — The polysomnography (referred to as type I) allows assessing several sleep physiologic parameters (eg, EEG, electrooculogram, electromyogram, electrocardiogram, airflow, respiratory effort, oxygen saturation), whereas audio-video recording enables documenting tooth-grinding sounds and distinguishing between rhythmic masticatory muscle activity (RMMA) and orofacial (eg, swallowing) and other muscular activity (eg, head movements) during sleep. Based on the RMMA index (number of episodes per hour of sleep), sleep bruxism is diagnosed when RMMA episodes are greater than or equal to 2 (low-frequency SB, mild bruxism) or RMMA episodes are greater than or equal to 4 (high-frequency SB, severe bruxism)

SUMMARY:
This case-control study will evaluates the association between the definitive sleep bruxism diagnosis by gold-standard polysomnography examination obtained at Pelotas Sleep Institute and the sociodemographic, occupational, clinical conditions, sleep quality, sleep structure and Epworth sleepiness scale variables.

DETAILED DESCRIPTION:
Currently, as sleep and awake bruxism are generally considered as different behaviours observed during sleep and wakefulness, respectively, the single definition for bruxism is recommended be "retired" in favour of 2 separate definitions. In this sense, the sleep bruxism is a masticatory muscle activity during sleep that is characterised as rhythmic (phasic) or non-rhythmic (tonic) and is not a movement disorder or a sleep disorder in otherwise healthy individuals .The diagnosis of sleep bruxism often is challenging and despite the use of questionnaires, clinical exams and portable devices, based on current knowledge, the polysomnography with audio-video recordings emerges as the gold-standard criteria for a definite sleep bruxism diagnosis.

Included on the questionnaire there is a registration form, which contains: Sociodemographic: self-reported ethnicity, marital status, education level; Occupational: individuals were asked about work outside home, working hours; Clinical condition: body mass index, smoking; alcohol consumption; use of sleeping pills.

Sleep Quality, was evaluated with the following questions: Sleep behavioral, how long does it take to sleep; restless sleep; nightmares; heartburn, obstructive sleep apnea by polysomnography. Bedtime, sleep time. Waking during the night, insomnia. Morning wake up, headache on waking; Lastly, Sleep structure data: sleep onset latency, rapid eye movement, sleep latency, wake time after sleep onset, total sleep time, sleep efficiency, non-rapid eye movement, sleep time in stages N1, N2, and N3, REM sleep time, arousal, arousal per hour, respiratory disturbance index, apnea-hypopnea index; and Epworth Sleepiness Scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 20 to 60 years) and elderly (aged > 60 years) (WHO-World Health Organization, 2015) who were undergone to polysomnography (PSG) at the Pelotas Sleep Institute (PSI);
* Adequate cognitive capacity to understand and answer the questionnaire.

Exclusion Criteria:

• Those which the participants were unable to answer the questionnaires and who presented a history of epilepsy that could interfere in the results of PSG.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are in the adult and elderly age group and who seek or are referred to the Pelotas Sleep Institute for polysomnography in the period from January 2015 to December 2017 were assessed.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Sleep Bruxism | 4 months
  Patients included in the study received diagnosis of SB by polysomnography exams. The data were obtained from polysomnography records in which masseter electromyography (EMG) burst was detected based on a predefined EMG threshold (20% of maximal voluntary tooth clenching task). Right masseter EMG bursts exceeding 0.25 second in duration were selected for oromotor activity scoring according to published criteria. Oromotor episodes separated by 3-second intervals were recognized as rhythmic masticatory muscle activity (RMMA) if they corresponded to 1 of the 3 following patterns: phasic (3 or more EMG bursts, each lasting 0.25 to 2 seconds), tonic (1 EMG burst lasting more than 2 seconds), or mixed (both burst types) episodes. EMG bursts were considered within the same RMMA episode if the interval between them was shorter than 2 seconds. Participants had SB diagnosed by polysomnography (PSG) if the RMMA index was greater than 2 episodes per hour of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Lavigne GJ, Rompre PH, Montplaisir JY. Sleep bruxism: validity of clinical research diagnostic criteria in a controlled polysomnographic study. J Dent Res. 1996 Jan;75(1):546-52. doi: 10.1177/00220345960750010601. PMID 8655758
- [Background] Casett E, Reus JC, Stuginski-Barbosa J, Porporatti AL, Carra MC, Peres MA, de Luca Canto G, Manfredini D. Validity of different tools to assess sleep bruxism: a meta-analysis. J Oral Rehabil. 2017 Sep;44(9):722-734. doi: 10.1111/joor.12520. Epub 2017 Jun 5. PMID 28477392
- [Background] Palinkas M, De Luca Canto G, Rodrigues LA, Bataglion C, Siessere S, Semprini M, Regalo SC. Comparative Capabilities of Clinical Assessment, Diagnostic Criteria, and Polysomnography in Detecting Sleep Bruxism. J Clin Sleep Med. 2015 Nov 15;11(11):1319-25. doi: 10.5664/jcsm.5196. PMID 26235152